- The effect of per oral immunotherapy treatment in severe IgE mediated egg, milk and nut allergy in adults.

NCT01822353

- The effect of per oral immunotherapy treatment in severe IgE mediated egg, milk and nut allergy in adults.

NCT01822353

## 3. Statistical methods

Frequencies, means, medians, proportions and standard deviations are calculated for all the data. Pairwise IgE results, methacholine challenge test results are analyzed using the nonparametric Wilcoxon signed rank test. Comparison of groups is done with chi square test and comparison of other continuous variables is done with t-test or with Mann-Whitney test. A p-value of less than 0.05 is considered statistically significant. The analyses will be performed using the SPSS 19.0 software package (SPSS Inc., Chicago, IL, USA).